CLINICAL TRIAL: NCT02536378
Title: POST-APPROVAL STUDY of TRANSCAROTID ARTERY REVASCULARIZATION in PATIENTS With SIGNIFICANT CAROTID ARTERY DISEASE. The ROADSTER 2 Study.
Brief Title: POST-APPROVAL STUDY of TRANSCAROTID ARTERY REVASCULARIZATION in PATIENTS With SIGNIFICANT CAROTID ARTERY DISEASE
Status: Completed | Type: Observational
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: SRM-2015-02
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The ROADSTER 2 Study is intended to evaluate real world usage of the ENROUTE Transcarotid Stent when used with the ENROUTE Transcarotid Neuroprotection System by physicians of varying experience with the transcarotid technique.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient must meet one of the following criteria regarding neurological symptom status and degree of stenosis:

   Symptomatic: Stenosis must be >50% as determined by an angiogram and the patient has a history of stroke (minor or non-disabling; NIHSS ≤4 or mRS ≤2), TIA and/or amaurosis fugax within 180 days of the procedure procedure ipsilateral to the carotid artery to be stented.

   OR Asymptomatic: Stenosis must be >80% as determined by angiogram without any neurological symptoms within the prior 180 days.
2. Target vessel must meet all requirements for ENROUTE Transcarotid Neuroprotection System and ENROUTE Stent System (refer to IFU for requirements).
3. Patient has a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA).
4. Patient is ≥18 years of age.
5. Patient understands the nature of the procedure and has provided a signed informed consent using a form that has been reviewed and approved by the Institutional Review Board/Ethics Committee of the respective clinical site prior to the procedure. This will be obtained prior to participation in the study.
6. Patient is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.
7. Patient must have a life expectancy ≥ 3 years at the time of the index procedure without contingencies related to other medical, surgical or endovascular intervention.
8. Patient meets at least one of the surgical high-risk criteria listed below.

Anatomic High Risk Inclusion Criteria:

A. Contralateral carotid artery occlusion B. Tandem stenoses >70% C. High cervical carotid artery stenosis D. Restenosis after carotid endarterectomy E. Bilateral carotid artery stenosis requiring treatment within 30 days after index treatment.

F. Hostile Necks which the Investigator deems safe for transcarotid access including but not limited to:

I. Prior neck irradiation II. Radical neck dissection III. Cervical spine immobility

Clinical High Risk Inclusion Criteria:

G. Patient is > 75 years of age H. Patient has > 2-vessel coronary artery disease and history of angina of any severity I. Patient has a history of angina

* Canadian Cardiovascular Society (CCS) angina class 3 or 4 or
* unstable angina

J. Patient has congestive heart failure (CHF) - New York Heart Association (NYHA)

* Functional Class III or IV

K. Patient has known severe left ventricular dysfunction

* LVEF <30%.

L. Patient has had a myocardial infarction > 72 hours and < 6 weeks prior to procedure.

M. Patient has severe pulmonary disease (COPD) with either:

* FEV1 <50% predicted or
* chronic oxygen therapy or
* resting PO2 of <60 mmHg (room air)

N. Patient has permanent contralateral cranial nerve injury O. Patient has chronic renal insufficiency (serum creatinine > 2.5 mg/dL).

REMINDER: The following is a list of anatomical considerations that are not suitable for transfemoral CAS with distal protection that are NOT contraindications for enrollment in the ROADSTER 2 Study including but not limited to:

I. TypeII, III, or Bovine arch II. Arch atheroma or calcification III. Atheroma of the great vessel origins IV. Tortuous distal ICA V. Tortuous or occluded iliofemoral segments VI. Occluded aortoiliac segments

EXCLUSION CRITERIA:

Each potential patient must be screened to ensure that they do not meet any of the following exclusion criteria. This screening is to be based on known medical history and data available at the time of eligibility determination and enrollment.

1. Patient has an alternative source of cerebral embolus, including but not limited to:

   1. Patient has chronic atrial fibrillation.
   2. Patient has had any episode of paroxysmal atrial fibrillation within the past 6 months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation.
   3. Knowledge of cardiac sources of emboli. e.g. left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma).
   4. Recently (<60 days) implanted heart valve (either surgically or endovascularly), which is a known source of emboli as confirmed on echocardiogram.
   5. Abnormal angiographic findings: ipsilateral intracranial or extracranial arterial stenosis (as determined by angiography or CTA/MRA ≤ 6 months prior to index procedure) greater in severity than the lesion to be treated, cerebral aneurysm > 5 mm, AVM (arteriovenous malformation) of the cerebral vasculature, or other abnormal angiographic findings.
2. Patient has a history of spontaneous intracranial hemorrhage within the past 12 months, or has had a recent (<7 days) stroke of sufficient size (on CT or MRI) to place him or her at risk of hemorrhagic conversion during the procedure.
3. Patient had hemorrhagic transformation of an ischemic stroke within the past 60 days.
4. Patient with a history of major stroke attributable to either carotid artery (CVA or retinal embolus) with major neurological deficit (NIHSS ≥ 5 OR mRS ≥ 3) likely to confound study endpoints within 1 month of index procedure.
5. Patient has an intracranial tumor.
6. Patient has an evolving stroke.
7. Patient has neurologic illnesses within the past two years characterized by fleeting or fixed neurologic deficit which cannot be distinguished from TIA or stroke, including but not limited to: moderate to severe dementia, partial or secondarily generalized seizures, complicated or classic migraine, tumor or other space-occupying brain lesions, subdural hematoma, cerebral contusion or other post-traumatic lesions, intracranial infection, demyelinating disease, or intracranial hemorrhage).
8. Patient has had a TIA or amaurosis fugax within 48 hrs prior to the procedure.
9. Patient has an isolated hemisphere.
10. Patient had or will have CABG, endovascular stent procedure, valve intervention or vascular surgery within 30 days before or after the intervention.
11. Myocardial Infarction within 72 hours prior to the intervention.
12. Presence of a previous placed intravascular stent in target vessel or ipsilateral CCA or significant CCA inflow lesion.
13. Occlusion or [Thrombolysis In Myocardial Infarction Trial (TIMI 0)] "string sign" >1cm of the ipsilateral common or internal carotid artery.
14. An intraluminal filling defect (defined as an endoluminal lucency surrounded by contrast, seen in multiple angiographic projections, in the absence of angiographic evidence of calcification) whether or not it is associated with an ulcerated target lesion.
15. Ostium of Common Carotid Artery (CCA) requires revascularization.
16. Patient has an open stoma in the neck.
17. Female patients who are pregnant or may become pregnant.
18. Patient has history of intolerance or allergic reaction to any of the study medications or stent materials (refer to stent IFU), including aspirin (ASA), ticlopidine, clopidogrel, statin or contrast media (that can't be pre medicated). Patients must be able to tolerate statins and a combination of ASA and ticlopidine or ASA and clopidogrel.
19. Patient must have a life expectancy <3 years without contingencies related to other medical, surgical, or interventional procedures as per the Wallaert Score and patients with primary, recurrent or metastatic malignancy who do not have independent assessment of life expectancy performed by the treating oncologist or an appropriate specialist other than the physician performing TCAR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atherosclerotic extracranial internal carotid stenosis (ICA) with or without involvement of the contiguous common artery (CCA) determined by duplex ultrasound, CT/CTA, MR/MRA or angiography to be:
  * Symptomatic: greater than or equal to 50% stenosis or
  * Asymptomatic: greater than or equal to 80% stenosis
Sampling Method: Non-Probability Sample
Enrollment: 692 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Kashyap, MD, Principal Investigator — University Hospital Case Medical Center Harrington Heart & Vascular Institute; Peter Schneider, MD, Principal Investigator — Kaiser Permanente
Locations (43):
- United States (41):
  - Peter Morton UCLA Medical Center, Los Angeles, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory Healthcare, Atlanta, Georgia
  - Kaiser Permanente, Hawaii, Honolulu, Hawaii
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Unity Point Health - Iowa Clinic, Des Moines, Iowa
  - Baptist Health Louisville, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Michigan Vascular Center, Flint, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Ct., Lebanon, New Hampshire
  - New Mexico, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Sisters of Charity Hospital, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - New Your Presbytarian - Weill Cornell, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook Medicine, Stony Brook, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - University Hospitals Case Medical Center and Case Western Reserve University School of Medicine, Cleveland, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC (University of Pittsburgh Medical Center), Pittsburgh, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Houston Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Sentara Vascular Specialists, Chesapeake, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Technical University Munich, Munich, Germany
- Hospital Quirónsalud Marbella, Marbella, Spain

REFERENCES:
- [Result] Alpaslan A, Wintermark M, Pinter L, Macdonald S, Ruedy R, Kolvenbach R. Transcarotid Artery Revascularization With Flow Reversal. J Endovasc Ther. 2017 Apr;24(2):265-270. doi: 10.1177/1526602817693607. Epub 2017 Feb 17. PMID 28335706
- [Derived] Chung J, Kumins NH, Smith J, Motaganahalli RL, Schneider PA, Kwolek CJ, Kashyap VS; ROADSTER Investigators. Physiologic risk factors increase risk of myocardial infarction with transcarotid artery revascularization in prospective trials. J Vasc Surg. 2023 Apr;77(4):1192-1198. doi: 10.1016/j.jvs.2022.12.013. Epub 2022 Dec 20. PMID 36563712
- [Derived] Kashyap VS, So KL, Schneider PA, Rathore R, Pham T, Motaganahalli RL, Massop DW, Foteh MI, Eckstein HH, Jim J, Leal Lorenzo JI, Melton JG. One-year outcomes after transcarotid artery revascularization (TCAR) in the ROADSTER 2 trial. J Vasc Surg. 2022 Aug;76(2):466-473.e1. doi: 10.1016/j.jvs.2022.03.872. Epub 2022 Apr 2. PMID 35381327
- [Derived] Kashyap VS, Schneider PA, Foteh M, Motaganahalli R, Shah R, Eckstein HH, Henao S, LaMuraglia G, Stoner MC, Melton J, Massop D, Hanover T, Titus J, Moore WS, Rodriguez-Carvajal R, Malas MB, Arko FR 3rd, Pierce D, Anain P, Oskin T; ROADSTER 2 Investigators*. Early Outcomes in the ROADSTER 2 Study of Transcarotid Artery Revascularization in Patients With Significant Carotid Artery Disease. Stroke. 2020 Sep;51(9):2620-2629. doi: 10.1161/STROKEAHA.120.030550. Epub 2020 Aug 19. PMID 32811386
- See also: Transcarotid Artery Revascularization With Flow Reversal: The PROOF Study — https://www.ncbi.nlm.nih.gov/pubmed/28335706

RESULTS

PARTICIPANT FLOW:
Groups:
- PP (Per Protocol): Patients who underwent the study procedure, independent of the success of the procedure and in the absence of major protocol deviations. The analysis of the PP population excludes those subjects for whom a major protocol deviation was identified by the CEC
- ITT (Intention to Treat): All patients who were enrolled in the pivotal phase of the study but had major protocol deviations
Period: Overall Study
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat)
Started | 632 | 60
Completed | 625 | 53
Not Completed | 7 | 7
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 1 | 2
Not completed — Patient refused further follow up | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- ITT (Intention to Treat): Patients who were enrolled in the pivotal phase of the study but had a major protocol deviation are included
- Total: Total of all reporting groups
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat) | Total
Number analyzed (Participants) | 632 | 60 | 692
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 104 | 9 | 113
  >=65 years | 528 | 51 | 579
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 19 | 223
  Male | 428 | 41 | 469
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 28 | 7 | 35
  Asian | 5 | 2 | 7
  Caucasian | 560 | 45 | 605
  Hispanic or Latino | 23 | 5 | 28
  Pacific Islander | 3 | 0 | 3
  Unknown/Other | 11 | 1 | 12
  Mixed Race | 2 | 0 | 2
Symptomatic Status [Count of Participants; unit: Participants]
  Asymptomatic | 466 | 46 | 512
  Symptomatic | 166 | 14 | 180
Height [Mean (Standard Deviation); unit: cm] | 170.3 (9.91) | 169.0 (11.8) | 170.2 (9.93)
Weight [Mean (Standard Deviation); unit: kg] | 81.5 (18.23) | 83.6 (18.72) | 81.7 (18.48)
High Surgical Risk Inclusion Criteria - Anatomic Risk Factors [Count of Participants; unit: Participants]
  Contralateral Carotid Artery Occlusion: Yes | 64 | 3 | 67
  Contralateral Carotid Artery Occlusion: No | 568 | 57 | 625
  Tandem Stenoses >70%: Yes | 10 | 3 | 13
  Tandem Stenoses >70%: No | 622 | 57 | 679
  High cervical carotid artery stenosis: Yes | 177 | 18 | 195
  High cervical carotid artery stenosis: No | 455 | 42 | 497
  Restenosis after carotid endarterectomy: Yes | 122 | 13 | 135
  Restenosis after carotid endarterectomy: No | 510 | 47 | 557
  Bilateral carotid artery stenosis req. treatment: Yes | 52 | 1 | 53
  Bilateral carotid artery stenosis req. treatment: No | 580 | 59 | 639
  Hostile necks safe for transcarotid access: Yes | 24 | 2 | 26
  Hostile necks safe for transcarotid access: No | 608 | 58 | 666
Medical History [Number; unit: Percentage of participants]
  Symptomatic | 26.3 | 23.3 | 26
  Male | 67.7 | 68.3 | 67.8
  Diabetes | 35 | 46.7 | 36
  Hypertension | 90.3 | 95.0 | 90.8
  History of Peripheral Artery Disease | 24.7 | 30.0 | 25.1
  History of Coronary Artery Disease | 14.6 | 10.0 | 14.2
  History of Angina | 2.1 | 0.0 | 1.9
  Congestive Heart Failure | 1.9 | 0.0 | 1.7
  Recent MI | 0.8 | 0.0 | 0.7
  Severe Pulmonary Disease | 2.8 | 1.7 | 2.7
  Dyslipidemia | 85.8 | 91.7 | 86.3
  History of Stroke | 15.7 | 23.3 | 16.4
  History of TIA | 16.1 | 15.0 | 16.0
  History of Amaurosis Fugax | 8.5 | 8.3 | 8.5
  Current Nicotine Use | 21.8 | 13.3 | 21.1
  Age ≥75 Years | 41.8 | 45.0 | 42.1
  Age ≥80 Years | 21.2 | 20.0 | 21.1
  Contralateral Carotid Occlusion | 10.1 | 5.0 | 9.7
  High Cervical Carotid Stenosis | 28 | 30.0 | 28.2
  Restenosis after CEA | 19.3 | 21.7 | 19.5
  Bilateral Stenosis Requiring Treatment | 8.2 | 1.7 | 7.7
  Hostile Neck Safe for Transcarotid Access | 3.8 | 3.3 | 3.8
  >2 Vessel Coronary Disease | 14.6 | 10.0 | 14.2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural Success
Description: Procedural success is defined as acute device success (successful insertion of the ENROUTE NPS and establishment of flow reversal), technical success (deployment of interventional tools) and the absence of a major adverse events (hierarchical stroke/death/myocardial infarction) through 30 days.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Groups:
- ITT (Intention to Treat): All patients who were enrolled in the pivotal phase of the study, including patients with major protocol deviations
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat)
Number analyzed (Participants) | 632 | 692
Participants | 630 | 690

2. Secondary Outcome: Number of Participants Experiencing Major Adverse Event
Description: Secondary endpoints include the 30-day rate of hierarchical stroke, death or myocardial infarction, the rate of hierarchical stroke, death or myocardial infarction by symptom status, the rate of cardiac death and the rate of neurological death.
Time Frame: 30 days
Population: 30 day Major Adverse Events as adjudicated by CEC
Measure: Number; unit: Major Adverse Events
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat)
Number analyzed (Participants) | 632 | 692
Major Adverse Events
  Death | 1 | 3
  Stroke | 4 | 13
  Myocardial Infarction | 6 | 6

3. Secondary Outcome: Number of Participants With Acute Device Success
Description: Acute device success is defined as the ability to insert the device, establish flow reversal, and remove the device
Time Frame: 2 hours (periprocedural)
Population: 2 enrolled patients were withdrawn by the Investigator
Measure: Count of Participants; unit: Participants
Groups:
- ITT (Intention to Treat): All patients who were enrolled in the pivotal phase of the study in which a major protocol deviation was identified by the CEC.
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat)
Number analyzed (Participants) | 632 | 692
Participants | 630 | 690

4. Secondary Outcome: Number of Participants With Technical Success
Description: Technical success is defined as acute device success plus the ability to deliver interventional tools
Time Frame: 2 hours (periprocedural)
Measure: Count of Participants; unit: Participants
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat)
Number analyzed (Participants) | 632 | 692
Participants | 630 | 690

5. Secondary Outcome: Number of Participants in Which a Cranial Nerve Injury Occurred
Description: Rate of cranial nerve injury suspected to be caused by surgical procedure and adjudicated by CEC.
Time Frame: 90 days (extended follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat)
Number analyzed (Participants) | 632 | 692
Participants | 8 | 10

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the life of the study: 3 years, 6 months
Description: Major adverse events, cranial nerve injuries, device related, and unanticipated adverse device effect event data were collected through 30 day follow-up period and recorded on the Adverse Event CRF. The Investigator or Coordinator determined whether an adverse event occurred
  Major Adverse Events were defined in this study as stroke, death, or myocardial infarction as adjudicated by Clinical Events Committee.
  Other Adverse Events (non-serious) were not collected or assessed for this study
Arm/Group | PP (Per Protocol) | ITT (Intention to Treat)
All-Cause Mortality (participants affected / at risk) | 1/632 | 3/692
Serious Adverse Events (participants affected / at risk) | 27/632 | 14/692
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PP (Per Protocol) (N=632) | ITT (Intention to Treat) (N=692)
Cranial Nerve Injury (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10) — Injury to cranial nerves in the vicinity of the treated carotid artery that has not resolved by one month after the initial procedure.
Death - Neurological (Nervous system disorders) | 0 (0) | 2 (2) — Death due to stroke or other neurologic cause
Death - Other (General disorders) | 1 (1) | 1 (1) — Death that cannot be attributed to neurologic or cardiac causes
Myocardial Infarction (Cardiac disorders) | 6 (6) | 7 (7) — Myocardial ischemia with elevation of cardiac enzymes (CK-MB or troponin) to a value 2 or more times the individual clinical center's laboratory upper limit of normal
NPS Device Related Event (Surgical and medical procedures) | 2 (2) | 2 (2) — Includes dissection and any vascular complication that may be attributed to the procedure or devices
Stroke - Contralateral (Nervous system disorders) | 1 (1) | 1 (1) — A neurological deficit attributed to an acute focal injury of the central nervous system contralateral to the vessel being stented.
Stroke - Ipsilateral (Nervous system disorders) | 3 (3) | 14 (14) — A neurological deficit attributed to an acute focal injury of the central nervous system ipsilateral to the vessel being stented
Possibly NPS/Stent device related event (Surgical and medical procedures) | 5 (5) | 7 (7) — Includes dissection, and any vascular complication that may be attributed to the procedure or devices
Stent Device Related Event (Surgical and medical procedures) | 1 (1) | 1 (1) — Includes thrombus formation, and any vascular complication that may be attributed to the procedure or devices

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02536378/Prot_SAP_000.pdf